CLINICAL TRIAL: NCT03995901
Title: A Randomized, Controlled, Multi-center, Safety and Efficacy Study of FCR001 Cell-based Therapy Relative to a Tacrolimus and Mycophenolate-based Regimen in de Novo Living Donor Renal Transplant Recipients, and Safety in FCR001 Donors
Brief Title: A Safety and Efficacy Study of FCR001 vs Standard of Care in de Novo Living Donor Kidney Transplantation
Acronym: FREEDOM-1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Talaris decided to discontinue living donor kidney transplant development program
Sponsor: Talaris Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FCR001A2301
Record Dates: First submitted 2019-06-13; First posted 2019-06-24 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Transplanted Organ Rejection
Keywords: Kidney Transplant; Stem cell therapy; Anti-rejection medications; Living donor kidney transplant; Immune tolerance; Immunosuppression; Immunosuppressive medication; Organ transplant rejection
MeSH Terms: interventions — Cell- and Tissue-Based Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FCR001 (Experimental): FCR001 is a cryopreserved allogeneic stem cell therapy derived from mobilized peripheral blood of the kidney donor that is delivered as a single dose with a non- myeloablative conditioning regimen. FCR001 contains the donor's CD34+ cells, facilitating cells, and αβ T cells.
  Interventions: Biological: FCR001
- Control (No Intervention): Standard induction therapy followed by a maintenance regimen of tacrolimus, mycophenolate, and +/- corticosteroids after kidney transplant.
  Control donors are not followed beyond randomization.

INTERVENTIONS:
Biological: FCR001 — FCR001 is a cryopreserved allogeneic stem cell therapy derived from mobilized peripheral blood of the kidney donor that is delivered as a single dose with a non- myeloablative conditioning regimen. FCR001 contains the donor's CD34+ cells, facilitating cells, and αβ T cells.
  Other Names: Cell based therapy; Allogeneic stem cell transplant
  Arms: FCR001

SUMMARY:
A randomized controlled study to evaluate the safety, efficacy, and overall benefit of FCR001 cell therapy in de novo living donor renal transplantation.

DETAILED DESCRIPTION:
The purpose of this randomized (2:1) controlled study is to evaluate the safety, efficacy and overall benefit of FCR001 cell therapy in first or second de novo living donor renal transplantation relative to a standard-of-care control immunosuppression regimen of antibody induction, tacrolimus, mycophenolate, and corticosteroids.

ELIGIBILITY:
Main Inclusion Criteria:

* Recipient age ≥18 years.
* Donor age ≥18 and ≤60 years at time of signing informed consent.
* Recipients of a first or second living donor kidney transplant
* Donor willing to undergo mobilization, apheresis and 12-month safety follow-up and meet all local standard eligibility criteria to donate stem cells for allogeneic transplantation.
* Recipient meets all local standard eligibility criteria for allogeneic stem cell transplant.
* Donors must be deemed eligible as per the requirements of 21CFR1271.

Main Recipient and Donor Exclusion Criteria:

* Recipient and donor who are identical twins.
* Recipient or donor with history of malignancy or premalignant syndrome (e.g., myelodysplastic syndrome, monoclonal gammopathy of renal significance [MGRS], monoclonal gammopathy of unknown significance [MGUS]) of any organ system (other than localized basal cell carcinoma of the skin or in-situ cervical cancer), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
* Recipient or donor with known bone marrow aplasia.

Main Recipient-only Exclusion Criteria:

* Multi-organ or stem cell transplant recipient.
* Calculated panel reactive antibodies >80%.
* Recipient is blood type ABO incompatible with donor.
* Presence of donor-specific antibodies (DSA) (positive result) at any time pre-transplant.
* Recipient who is human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) positive.
* Recipient with any baseline condition requiring or anticipated will require chronic or intermittent use of systemic steroids or other IS (eg, autoimmune disease, asthma) throughout the course of the study.
* Recipient with a BMI < 18 or > 35 kg/m2.
* Recipient requiring systemic anticoagulation, (eg, for hyper-coagulation disorders, deep vein thrombosis, atrial fibrillation) that cannot be temporarily interrupted which would preclude renal biopsy.

Main Donor-only Exclusion Criteria:

* Biologically unrelated (i.e., no genetic relationship) female donor transplant to male recipient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2023-02-16 (Actual)

PRIMARY OUTCOMES:
Proportion of FCR001 recipients who are free from immunosuppression (IS), without biopsy proven acute rejection (BPAR) at 24 months post-transplant | 24 months post-transplant
  Free from IS is defined as not taking any immunosuppression medications and not having to take immunosuppression medications since their withdrawal.
  Biopsy proven acute rejection is defined as Grade ≥1A according to the Banff 2017 Classification of Antibody-Medicated Rejection and T Cell-Mediated Rejection in Renal Allografts (Haas et al 2018).

SECONDARY OUTCOMES:
Change in renal function by Modification of Diet in Renal Disease (MDRD4) from post-transplant baseline (Month 1) to Month 24 in FCR001 recipients | 24 months post-transplant
Proportion of FCR001 recipients free from IS, without BPAR, at Month 36 and 60 | Month 36 and 60 post transplant
Allograft function (eGFR by MDRD4) and change in eGFR from Month 1 to Month 24, 36, and Month 60, by treatment | Month 1 (post-transplant) to Month 24, 36, and Month 60
Slope and difference in slope of estimated glomerular filtration rate (eGFR) by Modification of Diet in Renal Disease (MDRD4) over time to Month 24, 36, and 60, by treatment | Month 24, 36, and 60
Allograft function (eGFR) and change in renal allograft function from Month 1 to Months 24, 36 and 60 by treatment group, using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula | Month 1 (post transplant) to Month 24, 36, and Month 60
Time to the event for the composite of BPAR, graft loss, death or lost to follow-up and for each component, by treatment group | Month 1 (post transplant) to Month 6, 12, 24, 36, and 60
Incidence of composite endpoint of BPAR, graft loss or death, by treatment group | Months 12, 24, 36 and 60
Incidence of composite endpoint of BPAR, graft loss, or death and lost to follow-up, by treatment group | Months 12, 24, 36 and 60
Incidence of BPAR and treated BPAR by severity, type, and steroid-resistance, by treatment group | Months 12, 24, 36 and 60
Incidence of acute rejection | Months 12, 24, 36 and 60
Incidence of de novo donor-specific antibodies | Months 12, 24, 36 and 60
Incidence or worsening of abnormal histologic findings of cellular or antibody-mediated chronic rejection, chronic glomerulopathy, tubular atrophy and interstitial fibrosis, C4d, calcineurin inhibitor induced damage, disease recurrence, BK nephropathy | Months 12, 24, 36 and 60
Incidence of renal replacement therapy by treatment group | Months 12, 24, 36 and 60
Incidence of BPAR or eGFR <50 mL/min by treatment group | Months 12, 24, 36 and 60
Categorical distribution of eGFR according to chronic kidney disease CKD staging classification by treatment | Months 12, 24, 36 and 60
Incidence and severity of adverse events (AEs; including infections), serious adverse events (SAEs) and AEs leading to study and/or regimen discontinuation | Months 12, 24, 36 and 60
Incidence of BK viremia, viruria, infection, and nephropathy by treatment | Months 12, 24, 36 and 60
Incidence of the adverse events of special interest (proteinuria, neurotoxicity, anemia, diabetes, hypertension, dyslipidemia, opportunistic infections, major adverse cardiovascular events, and malignancies | Months 12, 24, 36 and 60
Urinary protein and albumin excretion, estimated by urinary protein/creatinine and urinary albumin/creatinine ratios by treatment group | Months 12, 24, 36 and 60
Subject quality of life according to 36-Item Short Form Health Survey (SF-36) will be analyzed descriptively by treatment group | Months 12, 24, 36 and 60
Subject quality of life according to End-Stage Renal Disease Symptom Checklist (ESRD-SCL) will be analyzed descriptively by treatment group | Months 12, 24, 36 and 60
Incidence and duration of hospitalization and readmission, according to type of ward/unit | Months 12, 24, 36 and 60
iBox predicted allograft survival | Months 12 and 24 post-transplant
Graft and patient survival and eGFR in FCR001 recipients who are only transiently chimeric | Month 24, 36, and 60
To describe the incidence and severity of AEs (including infections) and SAEs among FCR001 donors | Month 24, 36, and 60
Incidence of acute rejection, death, renal graft loss, and lost to follow-up between FCR001 recipients who did not achieve durable chimerism or the ability to wean or remain off immunosuppression vs. the control arm | Month 24, 36, and 60
The incidence of autologous infusions in FCR001 recipients | Month 6, 12, 24, 36, and 60
The incidence of engraftment syndrome in FCR001 recipients | Month 6, 12, 24, 36, and 60
The incidence of blood component transfusions in FCR001 recipients | Month 6, 12, 24, 36, and 60
The time to neutrophil and platelet recovery in FCR001 recipients | Month 6, 12, 24, 36, and 60
The incidence of acute and chronic Graft versus Host Disease (GvHD) in FCR001 recipients will be described | Month 6, 12, 24, 36, and 60
The incidence of donor chimerism and level of chimerism by study visit in FCR001 recipients will be described | Month 6, 12, 24, 36, and 60
The correlation of donor chimerism with freedom from IS)in FCR001 recipients will be described | Month 6, 12, 24, 36, and 60

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Mayo Clinic, Phoenix, Arizona
  - Scripps Clinic, La Jolla, California
  - University of California, San Francisco, San Francisco, California
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Mayo Clinic, Jacksonville, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - The University of Michigan Hospitals & Health System, Ann Arbor, Michigan
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - New York-Presbyterian/Weill Cornell, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Baylor University Medical Center, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No